CLINICAL TRIAL: NCT02849951
Title: A Randomized, Double-blind, Placebo-controlled Study of the Efficacy and Safety of a 12-week Add-on Treatment With LT-02 vs. Placebo in Subjects With Ulcerative Colitis Refractory to Standard Treatment With Mesalamine
Brief Title: A Study to Investigate the Safety and Efficacy of LT-02 in Patients With Mesalamine Refractory Ulcerative Colitis (UC)
Acronym: PROTECT-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: LT-02 did not appear to help induce remission of UC
Sponsor: Prometheus Laboratories (Industry)
Collaborators: Nestlé Health Science Spain (Industry); Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16GI01
Record Dates: First submitted 2016-07-26; First posted 2016-07-29 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Ulcerative Colitis
Keywords: Colitis; Colitis, Ulcerative; Ulcer; Colonic Diseases; Digestive System Diseases; Gastroenteritis; Gastrointestinal Diseases; Inflammatory Bowel Diseases; Intestinal Diseases; Pathologic Processes; Mesalamine
MeSH Terms: conditions — Colitis, Ulcerative; Colitis; Ulcer; Colonic Diseases; Digestive System Diseases; Gastroenteritis; Gastrointestinal Diseases; Inflammatory Bowel Diseases; Intestinal Diseases; Pathologic Processes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LT-02 (Experimental): 1.6 g PC in LT-02 BID
  Interventions: Drug: LT-02
- LT-02 Placebo (Placebo Comparator): 0 g PC in LT-02 Placebo BID
  Interventions: Drug: LT-02 Placebo

INTERVENTIONS:
Drug: LT-02 — 12-weeks of 1.6 g BID delayed-release phosphatidylcholine (LT-02)
  Arms: LT-02
Drug: LT-02 Placebo — 12-weeks of 0 g BID delayed-release phosphatidylcholine (LT-02) placebo
  Arms: LT-02 Placebo

SUMMARY:
The purpose of this study is to determine whether Phosphatidylcholine (LT-02) add on treatment is effective and safe for the induction of remission in ulcerative colitis patients refractory to standard treatment with mesalamine

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study to assess the efficacy and safety of LT-02 (delayed release phosphatidylcholine granules; administered orally via 1.6 g BID for up to 12 weeks) in subjects with active ulcerative colitis who are refractory to a standard dose of oral mesalamine therapy. Refractory to mesalamine is defined as active disease despite receiving at least ≥ 2.4g mesalamine (or equivalent dose) for at least 8 weeks with or without rectal 5-ASA.

ELIGIBILITY:
Key Inclusion Criteria:

1. Established diagnosis of ulcerative colitis (UC), based on clinical history, exclusion of infectious causes, and characteristic endoscopic and histologic findings.
2. Active UC with disease confirmed by endoscopy findings and confirmed by central reader.
3. A modified Mayo Score 4-10, and with a centrally read endoscopy score activity of ≥ 2 points.
4. Mesalamine (5-ASA) refractory.

Exclusion Criteria:

1. Diagnosis of Crohn's disease, indeterminate colitis, ischemic colitis, radiation colitis, microscopic colitis (i.e., collagenous colitis and lymphocytic colitis), diverticular disease associated colitis,
2. Toxic megacolon or fulminant colitis,
3. Prior colon resection,
4. Evidence of infectious colitis (e.g., pathogenic bacteria or Clostridium difficile infection) at screening,
5. Known celiac disease
6. Other inflammatory or bleeding disorders of the colon and intestine, or diseases what may cause diarrhea or gastrointestinal bleeding
7. History or presence of ischemic heart disease, myocardial infarction, peripheral arterial disease, ischemic stroke, or transient ischemic attack,
8. Subjects with known hypersensitivity to soy,
9. Treatment with methotrexate, azathioprine, 6-mercaptopurine TNF-alpha-antagonists, vedolizumab or certolizumab pegol, tacrolimus, or anti-integrin therapy within last 8 weeks prior to screening,
10. Treatment with any (topical or systemic) corticosteroid formulation for the treatment of IBD within last 7 days prior to endoscopy,
11. Treatment with other investigational drug within last 8 weeks prior to screening,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-07; Primary Completion 2019-03 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical remission | 12 weeks
  The percentage of subjects in clinical remission using the abbreviated modified Mayo score

SECONDARY OUTCOMES:
Clinical response | 12 weeks
  Percentage of subjects with clinical response using the abbreviated modified Mayo score
Endoscopic response | 12 weeks
  Percentage of subjects with endoscopic response
Histological improvement | 12 weeks
  Percentage of subjects with histological improvement
Endoscopic remission | 12 weeks
  Percentage of subjects with endoscopic remission
Mucosal healing | 12 weeks
  Percentage of subjects with mucosal healing
Quality of life | 12 weeks
  Change in the subjects quality of life, using Inflammatory Bowel Disease Quality of Life Questionnaire (IBDQ)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Gordon, M.D., J.D., Study Director — Nestle Health Science, Medical Director
Locations (45):
- United States (45):
  - Prometheus Site 24, Phoenix, Arizona
  - Prometheus Site 10, Little Rock, Arkansas
  - Prometheus Site 15, Chula Vista, California
  - Prometheus Site 42, Lancaster, California
  - Prometheus Site 30, Oceanside, California
  - Prometheus Site 28, Rialto, California
  - Prometheus Site 2, Ventura, California
  - Prometheus Site 27, Lafayette, Colorado
  - Prometheus Site 45, Lone Tree, Colorado
  - Prometheus Site 35, Clearwater, Florida
  - Prometheus Site 17, Fort Lauderdale, Florida
  - Prometheus Site 55, Hialeah, Florida
  - Prometheus Site 8, Naples, Florida
  - Prometheus Site 13, Naples, Florida
  - Prometheus Site 36, Orlando, Florida
  - Prometheus Site 44, Orlando, Florida
  - Prometheus Site 37, Athens, Georgia
  - Prometheus Site 11, Decatur, Georgia
  - Prometheus Site 53, Chicago, Illinois
  - Prometheus Site 54, Hoffman Estates, Illinois
  - Prometheus Site 20, Topeka, Kansas
  - Prometheus Site 4, Shreveport, Louisiana
  - Prometheus Site 5, Chevy Chase, Maryland
  - Prometheus Research Site 1, Brockton, Massachusetts
  - Prometheus Site 6, Chesterfield, Michigan
  - Prometheus Site 51, Southfield, Michigan
  - Prometheus Site 48, Wyoming, Michigan
  - Prometheus Site 31, Plymouth, Minnesota
  - Prometheus Site 40, St Louis, Missouri
  - Prometheus Site 21, Lebanon, New Hampshire
  - Prometheus Site 22, Great Neck, New York
  - Prometheus Site 33, Poughkeepsie, New York
  - Prometheus Site 26, The Bronx, New York
  - Prometheus Site 41, Greenville, North Carolina
  - Prometheus Site 32, Kinston, North Carolina
  - Prometheus Site 43, Columbia, South Carolina
  - Prometheus Site 7, Rapid City, South Dakota
  - Prometheus Site 49, Houston, Texas
  - Prometheus Site 39, Humble, Texas
  - Prometheus Site 47, San Antonio, Texas
  - Prometheus Site 9, San Antonio, Texas
  - Prometheus Site 23, Orem, Utah
  - Prometheus Site 25, Salt Lake City, Utah
  - Prometheus Site 34, Charlottesville, Virginia
  - Prometheus Site 12, Richland, Washington

IPD SHARING:
Plan to Share IPD: No